CLINICAL TRIAL: NCT02051036
Title: A Pilot Study on Effectiveness and Safety of Moxibustion for Benign Prostate Hyperplasia With Lower Urinary Tract Syndrome
Brief Title: Moxibustion as an Adjuvant for Benign Prostatic Hyperplasia With Lower Urinary Tract Symptoms: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JUNGNAM KWON (Other)
Responsible Party: Sponsor-Investigator, JUNGNAM KWON, Professor, Korean Medicine Hospital of Pusan National University
Organization: Korean Medicine Hospital of Pusan National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NC1307
Record Dates: First submitted 2014-01-26; First posted 2014-01-31 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: BPH; Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy; Lower Urinary Tract Symptom
Keywords: moxibustion
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxibustion (Experimental): A series of moxibustion sessions within four weeks from the baseline with concurrent conventional medications for BPH.
  Interventions: Procedure: Moxibustion
- Waiting (No Intervention): Participants who will be allocated to waitlist will receive no moxibustion treatments throughout the 4 weeks while receiving other conventional managements for BPH. After 4 weeks, if participants choose to try the moxibustion treatment, the active acupuncture treatment will be provided for 4 weeks (2 sessions/week).

INTERVENTIONS:
Procedure: Moxibustion — In the moxibustion treatment group, 5 moxibustion points (bilateral SP6, LV3 and unilateral CV4) will be heated with indirect moxibustion (KangHwa, Korea).
  The moxa pillars will be removed when the patient feel hotness and require to remove them.
  The moxibustion will be conducted repeatedly unless patients feel the sense of heat up to seven times per session.
  Arms: Moxibustion

SUMMARY:
This study aims to explore the feasibility of moxibustion as a supplementary intervention and to assess the sample size for verifying the effectiveness and safety of integrative treatment involving moxibustion compared with conventional treatment for patients with benign prostate hyperplasia (BPH) accompanying moderate to severe lower urinary tract symptoms (LUTS).

DETAILED DESCRIPTION:
Patients who diagnosed as BPH with moderate to severe LUTS aged 20 to 80 years old will be divided into two groups, one is moxibustion plus conventional therapy group and the other is conventional therapy group.

Patients who belong to moxibustion plus conventional therapy group will be treated moxibustion for eight times by a Korean Medicine doctor with conventional therapy by a urologist.

Patients who belong to conventional therapy group will be treated with conventional therapy only, and they can receive moxibustion therapy after the clinical trial is finished.

IPSS, post void residual volume (PVR) and peak urine flow (Qmax) will be checked to evaluate the effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 20-80 years diagnosed with BPH with a prostate size over 20 gm
2. greater than or equal to eight score on IPSS
3. submit written consent
4. who can understand and answer IPSS.

Exclusion Criteria:

1. prostate or bladder malignancy
2. received herbal medication for lower urinary tract symptoms within 1 week
3. history of brain disease could cause urinary difficulty
4. having problems on answering IPSS due to cognitive impairment.
5. signs of acute urinary tract infection
6. Diabetic mellitus
7. Neurogenic bladder

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
International prostate symptom score (IPSS) at 4 weeks | four weeks after randomization

SECONDARY OUTCOMES:
Patient's global impression of change (PGIC) | visit 2,3,4,5,6,7,8, 9 in experimental group, visit 8,9 in control group
Maximum flow rate by uroflowmetry (Qmax) | Baseline and 12 weeks after randomization (both group)
Post-voiding residual urine in bladder (PVR) | Baseline and 12 weeks after randomization
Changing Process and Persistence of International Prostate Symptom Score (IPSS) | 2 weeks, 12 weeks after randomization
recruitment rate | 31-December-2015
compliance rate | after 12 weeks
  the attendance rate for treatment phase in integrative group, and for three major assessments (baseline, visit 9 and visit 10)
retention rate | after four weeks, after 12 weeks
  the ratio of 1) the number of patients who attend at the primary outcome assessment after four weeks versus the number of total participants, 2) the number of patients who attend the final assessment after 12 weeks versus the number of total participants, 3) the number of patients who returned the frequency-volume chart (FVC) versus the number of total participants.
adverse events | visit 1,2,3,4,5,6,7,8,9 in experimental group ; visit 1,8,9 in control group
  patients will be asked if adverse effects have developed

CONTACTS AND LOCATIONS:
Overall Officials: Jung Nam Kwon, PhD, Principal Investigator — Korean Medicine Hospital, Pusan National University
Locations (1):
- National Clinical Research Center, Korean Medicine Hospital, Pusan National University, Yangsa, Kyungsangnamdo, South Korea

REFERENCES:
- [Derived] Lee HY, Nam JK, Lee SD, Lee DH, Han JY, Yun YJ, Lee JH, Park HL, Park SH, Kwon JN. Moxibustion as an adjuvant for benign prostatic hyperplasia with lower urinary tract symptoms: a protocol for a parallel-group, randomised, controlled pilot trial. BMJ Open. 2015 Dec 11;5(12):e008338. doi: 10.1136/bmjopen-2015-008338. PMID 26656981